CLINICAL TRIAL: NCT06373263
Title: A Randomized Controlled Trial to Compare the Effectiveness of Dissemination Tools to Share Research Results With Patients - SPIN-CLEAR Trial #1
Brief Title: Evaluating Tools to Communicate Scleroderma Research Results to Patients - Trial #1
Acronym: SPIN-CLEAR #1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Senior Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-4165
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Scleroderma; Knowledge Translation; Dissemination Tools; E-Health; Intervention; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissemination tool (infographic) (Experimental): Infographic
  Interventions: Other: Dissemination Tool (Infographic)
- Plain-language summary (Active Comparator): Plain-language summary
  Interventions: Other: Plain-language summary

INTERVENTIONS:
Other: Plain-language summary — Participants will receive information about a research study via a plain-language summary. The comparator will be a plain-language summary, since plain-language summaries are commonly used and more easily developed than other tools. The summary will be designed based on Canadian government and other key recommendations, including from the Cochrane Collaboration. It will include Background and Objectives, Methods, Results, Limitations, and Key Message for Patients sections and include information on how evidence informs knowledge or health care options. Abstract will be < 500 words long and use short, positive, active-voice sentence structures and everyday words. Reading level will be between 8th and 9th grade based on Flesch-Kincaid Grade Level and readability score between 60 and 70 based on Flesch Reading Ease.
  Arms: Plain-language summary
Other: Dissemination Tool (Infographic) — The infographic will be developed based on key principles including clearly defining the audience and purpose; sharing a story, rather than just facts, with brief, clear messaging; highlighting main ideas; using an attractive title and images; and following principles of good graphic design.
  Arms: Dissemination tool (infographic)

SUMMARY:
Sharing research results with patients is required by ethical regulations. Yet, most researchers do not share results from their studies with patients. The investigators plan to conduct a series of randomized controlled trials among people with scleroderma, a rare autoimmune disease, in a large international cohort, to identify the most effective methods for communicating study results with patients.

The first trial in the series will compare a research dissemination tool (infographic) against a plain-language summary comparator. Participants will be randomly assigned to receive the dissemination tool or comparator. Study participants will rate communication tools for (1) information completeness; (2) understandability; and (3) ease of use of format. Our results can be used by researchers and patient organizations who disseminate research results so that they can tailor the way they disseminate results to patient needs.

DETAILED DESCRIPTION:
Background: Research ethics guidance mandates that study results be shared with participants, and CIHR's Knowledge Translation Strategy emphasizes dissemination to others with relevant lived experiences. Yet, most researchers do not share results with patients, and do not know which dissemination tools (e.g., lay summaries, infographics, podcasts) or tool features best facilitate effective communication. Only 3 randomized controlled trials (RCTs) have compared tool effectiveness, and none assessed which approaches work best for which patients. Comparative effectiveness trials are needed to build an evidence base to help us understand what tools are most effective for communicating different types of research to different patients. The investigators will use the multinational Scleroderma Patient-centered Intervention Network (SPIN) Cohort to conduct a series of RCTs to compare tools among people with systemic sclerosis, or scleroderma. The first trial in the series will compare a research dissemination tool (infographic) against a plain-language summary comparator.

Objectives: An effective tool must communicate information patients want to know, understandably, in an easy-to-use format. The trial will compare the effectiveness of an infographic and lay summary, overall and for patients with different sociodemographic or educational characteristics.

Primary Objectives: The first trial will compare tools based on (1) information completeness; (2) understandability; and (3) ease of use, as prioritized by our Patient Advisory Team.

Secondary Objectives: The investigators will evaluate comprehension of key aspects of disseminated research; likelihood that participants would enroll in a similar future study; and, for all primary and secondary outcomes, analyze effects by participant characteristics (e.g., age, country, language, education level, eHealth literacy).

Methods: Parallel-group RCT that will compare 2 tools (infographic and plain-language summary comparator. For this trial, SPIN patients and researchers will select systemic sclerosis research to disseminate. Tools will be developed by experienced tool developers, patients, and researchers. SPIN Cohort participants (N = 1,250 and growing) will be invited to enrol, and those enrolled will be randomized to a dissemination tool and complete outcomes. Response options will be 0 to 10 numerical rating scales (0 = strongly disagree, 10 = strongly agree). The primary analysis will be intention-to-treat, using a linear mixed effects model with multiple observations per participant (using the lmer function from the lme4 package in R).

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in SPIN Cohort, which requires a systemic sclerosis (SSc) classification by a site physician based on 2013 American College of Rheumatology/European League Against Rheumatism criteria, ≥18 years old, being fluent in English or French, and have completed one SPIN Cohort assessment in the last year.
2. External enrollment with patient-reported physician classification of SSc and age 18 or older.

Exclusion Criteria:

Patients not able to access or respond to questionnaires via the internet are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Completeness | Immediately Post-intervention (intervention and outcomes in one login - outcomes approx 30 min after randomization)
  "The information presented in the [tool - e.g., "infographic", "plain-language summary"] told me everything I wanted to know about the study".
  Response options = 0-10 numerical rating scales (0 = strongly disagree, 10 = strongly agree)
Understandability | Immediately Post-intervention (intervention and outcomes in one login - outcomes approx 30 min after randomization)
  "The information presented in the [tool] was easy to understand". Response options = 0-10 numerical rating scales (0 = strongly disagree, 10 = strongly agree)
Ease of use | Immediately Post-intervention (intervention and outcomes in one login - outcomes approx 30 min after randomization)
  "The [tool] was designed in a way that made it easy to use". Response options = 0-10 numerical rating scales (0 = strongly disagree, 10 = strongly agree)

SECONDARY OUTCOMES:
Please to have received results | Immediately Post-intervention (intervention and outcomes in one login - outcomes approx 30 min after randomization)
  "I am glad that I received the study results"); Response options = 0-10 numerical rating scales (0 = strongly disagree, 10 = strongly agree)
Intention to participate in future studies | Immediately Post-intervention (intervention and outcomes in one login - outcomes approx 30 min after randomization)
  "In the future, I would agree to participate in a similar study to the one presented in the [tool]". Response options = 0-10 numerical rating scales (0 = strongly disagree, 10 = strongly agree)
Open-ended items | Immediately Post-intervention (intervention and outcomes in one login - outcomes approx 30 min after randomization)
  "What did you like about the way the information was communicated?"; "What did you dislike about the way the information was communicated?"; "Do you have suggestions for improving how the information is communicated?"

IPD SHARING:
Plan to Share IPD: Yes
All data and materials will be provided upon reasonable requests to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after the collection of the primary outcome.
Access Criteria: Approval of proposed purpose for data access.

REFERENCES:
- [Background] Thombs BD, Adams C, Nassar EL, Carrier ME, Golberg M, Bharthi K, Wurz A, South A, Kwakkenbos L, Hoa S, Rice DB, Guillot G, Lawrie-Jones A, Sauve M, Bartlett SJ, Fortune C, Gietzen A, Gottesman K, Hudson M, Hummers LK, Malcarne VL, Mayes MD, Richard M, Stempel J, Wojeck RK, Blagrave K, Boruff JT, Cook V, Culos-Reed N, Frobert O, Gillies K, Granikov V, Hemkens LG, Jimenez EY, Kocher A, Leite C, Lim MAWT, Maltez N, Michalski J, Mieszczak T, Ndosi M, Pope J, Rannou F, Rozee K, Straus SE, Sydes MR, Thabane L, Varga J, Yap T, Zwarenstein M, Mouthon L, Benedetti A; SPIN Investigators. Master protocol for a series of cohort-based randomized controlled trials to test tools to communicate research results to study participants and others with relevant lived experience: the SPIN-CLEAR Trials. Trials. 2025 May 8;26(1):149. doi: 10.1186/s13063-025-08846-2. PMID 40340935